CLINICAL TRIAL: NCT02390141
Title: A Randomized, Placebo-controlled, Double-blind Trial of Multiple Ascending Doses of ZP4207 Administered to Healthy Volunteers to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ZP4207
Brief Title: Multiple Ascending Doses of ZP4207 Administered to HV to Evaluate the Safety, Tolerability, PKs and PDs of ZP4207
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZP4207-15007
Record Dates: First submitted 2015-02-28; First posted 2015-03-17 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ZP4207 (Experimental): Five multiple doses of ZP4207 in ascending doses
  Interventions: Drug: ZP4207
- Placebo (Placebo Comparator): Five multiple doses of corresponding placebo in ascending doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ZP4207
  Arms: ZP4207
Drug: Placebo
  Arms: Placebo

SUMMARY:
The trial is a single-centre, randomized, double-blind, phase 1b trial of multiple ascending doses of ZP4207 administered s.c. to healthy volunteers (HV) to evaluate the safety, tolerability, pharmakocinetic (PK) and pharmacodynamic (PD). Three cohorts of 8 subjects are planned. Within each cohort, the subjects will be randomly assigned to five repeated doses of ZP4207 or placebo in a 3:1 treatment allocation at trial site.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent obtained before any trial-related activities. (Trial-related activities are any procedures that would not have been performed during normal management of the subject).
2. Caucasian
3. Healthy male subject.
4. Age between 18 and 50 years, both inclusive.
5. Body weight between 70 and 90 kg (both inclusive)
6. Fasting plasma glucose concentration <= 100 mg/dL.
7. Considered generally healthy upon completion of medical history, physical examination, vital signs, ECG and analysis of laboratory safety variables, as judged by the Investigator.

Exclusion Criteria:

1. Known or suspected hypersensitivity to IMP or related products.
2. Previous participation in this trial. Participation is defined as randomized.
3. Previous treatment with ZP4207.
4. Receipt of any medicinal product in clinical development within 3 months before randomization in this trial.
5. History of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reaction.
6. Any history or presence of cancer except basal cell skin cancer or squamous cell skin cancer as judged by the Investigator.
7. Any history or presence of clinically relevant cardiovascular, pulmonary, respiratory, gastrointestinal, hepatic, renal, metabolic, endocrinological, haematological, dermatological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness as judged by the Investigator.
8. Any serious systemic infectious disease during four weeks prior to first dosing of the study drug, as judged by the Investigator.
9. Clinically significant abnormal values for haematology, biochemistry, coagulation, or urinalysis as judged by the Investigator.
10. Supine blood pressure at screening (after resting for at least 5 min in supine position) outside the ranges for systolic 95-140 mmHg blood pressure and for diastolic greater than 90 mmHg or symptoms and a heart rate at rest outside the range of 50-90 beats per minute (excluding white-coat hypertension; therefore, if a repeated measurement shows values within the range, the subject can be included in the trial).
11. Clinically significant abnormal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in supine position at screening, as judged by the Investigator.
12. Significant history of alcoholism or drug abuse as judged by the Investigator or consuming more than 21 units of alcohol per week (one unit of alcohol equals about 250 mL of beer, one glass of wine of 120 mL, or 20 mL spirits).
13. A positive result in the alcohol and/or urine drug screen at the screening visit.
14. Smoker (defined as a subject who is smoking more than 7 cigarettes or the equivalent per week) within the last month prior to screening and who is not able or willing to refrain from smoking and use of nicotine substitute products one day before first dosing and during the treatment period.
15. Positive to the screening test for Hepatitis Bs antigen or Hepatitis C antibodies and/or a positive result to the test for HIV-1/2 antibodies or HIV-1 antigen.
16. Any medication (prescription and non-prescription drugs) within 14 days before IMP administration, with the exception of paracetamol or acetylsalicylic acid for occasional use to treat acute pain.
17. Blood donation or blood loss of more than 500 mL within the last 3 months.
18. Mental incapacity, unwillingness, or language barriers precluding adequate understanding or co-operation.
19. Male who is sexually active and not surgically sterilized who and whose partner(s) is not using adequate contraceptive methods (adequate contraceptive measures include surgical sterilisation, hormonal intrauterine devices [coil], oral hormonal contraceptives, each in combination with spermicide-coated condoms), or who is not willing to refrain from sexual intercourse from the first dosing until 1 month after last dosing in the trial.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 28 days
  Number of participants with adverse events
Number of participants with adverse events | 28 days
  Changes or findings from baseline (normal ranges) in clinical safety laboratory assessments (including haematology, biochemistry, coagulation and urinalysis).
Number of participants with adverse events | 28 days
  Changes or findings from baseline in physical examination including Head, ears, eyes, nose, throat (HEENT), incl. thyroid gland
  * Heart, lung, chest
  * Abdomen
  * Skin and mucosae
  * Musculoskeletal system
  * Nervous system
  * Lymph node
  * Other findings)
Number of participants with adverse events | 28 days
  Changes or findings from baseline in vital signs (including systolic and diastolic blood pressure (mmHG) und heart rate (beats per minute), body temperature (°C), respiratory frequency (RF/min))
Number of participants with adverse events | 28 days
  Changes or findings from baseline in ECG Parameter (Heart rate, PQ, QRS, QT, QTcB)
Number of participants with adverse events | 28 days
  Findings in local tolerability by means of the following assessments:
  * spontaneous pain
  * pain on palpation
  * itching
  * redness
  * oedema
  * induration/infiltration
  * other
Number of participants with adverse events | 28 days
  Immunogenicity (Anti-ZP4207 Antibodies)

SECONDARY OUTCOMES:
Areas under the plasma concentration curve compared between first and last dosing | 5h
  Areas under the plasma concentration curve from 0 until 300min
Areas under the plasma concentration curve compared between first and last dosing | 5 h
  Areas under the plasma concentration curve from 0 until infinity
Plasma concentration curve compared between first and last dosing | 5 h
  Maximum observed ZP4207 concentration
Plasma concentration curve compared between first and last dosing | 5 h
  Time to maximum observed ZP4207 concentration
Plasma concentration curve compared between first and last dosing | 5 h
  Terminal elimination rate constant of ZP4207
Plasma concentration curve compared between first and last dosing | 5 h
  Terminal plasma elimination half-life calculated as t½=ln2/λz
Plasma concentration curve compared between first and last dosing | 5 h
  Apparent volume of distribution of ZP4207 based on plasma concentration values, estimated during the terminal phase
Pharmacokinetic endpoints compared between first and last dosing | 5 h
  Apparent plasma clearance rate of ZP4207 estimated during the terminal phase
Pharmacokinetic endpoints compared between first and last dosing | 5 h
  Mean residence time for plasma ZP4207
Pharmacodynamic endpoints compared between first and last dosing | 5 h
  Area under the plasma glucose curve from 0 until 300min
Pharmacodynamic endpoints compared between first and last dosing | 5 h
  Maximum observed plasma glucose concentration
Pharmacodynamic endpoints compared between first and last dosing | 5 h
  Time to maximum plasma glucose concentration
Pharmacodynamic endpoints compared between first and last dosing | 5 h
  Delta (time to increase) of glucose of 2 mmol/

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Hövelmann, MD, Principal Investigator — Profil GmbH
Locations (1):
- Profil GmbH, Neuss, Germany